CLINICAL TRIAL: NCT02911116
Title: A Pilot Study to Investigate Ustekinumab (STELARA) for the Treatment of Active Sight-Threatening Uveitis
Brief Title: Ustekinumab (STELARA) for the Treatment of Active Sight-Threatening Uveitis (STAR Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160169; 16-EI-0169
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2020-12

CONDITIONS: Uveitis
Keywords: Panuveitis; Intermediate Uveitis; Uveitis
MeSH Terms: conditions — Uveitis; Panuveitis; Uveitis, Intermediate | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Subcutaneous Only) (Experimental): Subcutaneous injections of Ustekinumab at baseline.
  Interventions: Drug: Ustekinumab
- Cohort 2 (IV and Subcutaneous) (Experimental): Initial IV infusion of ustekinumab at baseline followed by one subcutaneous injection at Week 8. In participants who demonstrate an allergic reaction to the baseline IV infusion, the second dose at Week 8 can also be administered as an IV infusion instead of a subcutaneous injection.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Subcutaneous Injection
Drug: Ustekinumab — Intravenous Infusion
  Arms: Cohort 2 (IV and Subcutaneous)

SUMMARY:
Background:

Uveitis is an inflammation of the eye that can cause vision loss. It is treated with medications and sometimes surgery. However, in many people, treatment does not always prevent loss of vision. A new medication, ustekinumab, reduces inflammation in patients with other inflammatory diseases. Therefore, it might be helpful in treatment of uveitis.

Objective:

To see if ustekinumab is safe and can help people with uveitis.

Eligibility:

People ages 18 and older with uveitis

Design:

Participants will be screened with:

Medical and eye disease history

Physical exam

Eye exam: The pupil is dilated with eye drops. A machine scans the back of the eye. Pictures are taken of the inside of the eye.

Blood and urine tests

Tuberculosis test

Participants will have 6 clinic visits over 28 weeks. Visits lasts 2-3 hours and include:

* Medical and eye disease history
* Physical and eye exams
* Blood and urine tests
* Fluorescein angiography: A needle guides a thin plastic tube into an arm vein. A dye is injected into the tube. The dye travels through the veins up to the blood vessels in the eyes. A camera takes pictures of the dye as it flows through the blood vessels in the eyes.
* Cohort 1 - Ustekinumab injections at Weeks 0, 4, and 8: The injection is under the skin of the upper arm, leg, or abdomen.

Participants will have their uveitis monitored and receive standard uveitis care during the study.

* Cohort 2 - Ustekinumab injections via intravenous (IV) injection at first visit, followed by a single 90 mg injection of ustekinumab under the skin of the upper arm, leg or abdomen. For the IV injection a needle will be used to guide a thin plastic tube (catheter) into one of the arm veins. The needle will be removed, leaving only the catheter in the vein.

DETAILED DESCRIPTION:
Objective: Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects and many patients continue to experience disease flare-ups. Ustekinumab is a human IL-12 and -23 antagonist. The involvement of IL-12 and IL-23 in the pathophysiology of uveitis and other autoimmune diseases known to be associated with uveitis suggests that ustekinumab could be a potential treatment for uveitis. The study objective is to investigate the safety, tolerability and potential efficacy of ustekinumab as a possible treatment for active intermediate uveitis, posterior uveitis or panuveitis.

Study Population: The first cohort will consist of five participants with active intermediate uveitis, posterior uveitis or panuveitis who meet the inclusion criteria. The second cohort will include up to four participants with active intermediate uveitis, posterior uveitis or panuveitis who meet the inclusion criteria. Up to eleven participants may be enrolled, as up to two participants may be accrued in the second cohort to account for participants who withdraw from the study prior to Week 16.

Design: This is a prospective, non-randomized, uncontrolled, two-arm pilot study to evaluate of ustekinumab as a possible treatment for active intermediate uveitis, posterior uveitis or panuveitis. Five participants in the first cohort will receive a 90 mg subcutaneous (SC) injection of ustekinumab at baseline and a second and third injection at Week 4 and 8 for a total of 3 injections. For the second cohort, up to four participants will receive an initial high, weight-based dose of ustekinumab via intravenous (IV) injection (up to 55 kg, 260 mg (2 vials); greater than 55 kg to 85 kg, 390 mg (3 vials); greater than 85 kg, 520 mg (4 vials)), followed by a single 90 mg subcutaneous injection at Week 8. In participants who demonstrate allergic reaction to the first dose, the second dose can also be administered as IV infusion with pre-infusion desensitization instead of a subcutaneous injection as it allows better control on the rate of drug administration. Participants will continue in the study for a total of 28 weeks and will be able to receive standard of care after the first 16 weeks.

Outcome Measures: For each cohort, the primary outcome is the number of participants who experience treatment response by Week 16. Secondary outcomes for each cohort include changes in visual acuity, the number of participants who experience a recurrence, the number of days to recurrence, presence or extent of macular edema, the amount of retino-vascular leakage, changes in retinal thickening, the length of time to quiescence and the ability to taper concomitant immunosuppressive medications. Safety outcomes for each cohort include the number and severity of systemic and ocular toxicities and adverse events, the proportion of participants who experience vision loss of greater than or equal to 15 letters as measured by Electronic Visual Acuity (EVA) and the number of participants who experience a substantial rise in elevated intraocular pressure (IOP).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Participant has the ability to understand and sign the informed consent document.
2. Participant is 18 years of age or older.
3. Participant has negative purified protein derivative (PPD) or quantiferon testing done within three months prior to enrollment or had latent tuberculosis (TB) but has completed prophylactic anti-TB treatment.
4. Participant has active intermediate uveitis, posterior uveitis or panuveitis in at least one eye requiring systemic therapy. Active disease is defined as:

   * +1 or more vitreous haze (according to Standardization of Uveitis Nomenclature (SUN) criteria) AND/OR
   * Active chorioretinitis or leakage on Fluorescein angiography (FA)(that is in more than one quadrant) that requires treatment.
5. Participant has visual acuity in at least one eye of 20/400 or better.
6. Participant is willing and able to comply with the study procedures.
7. Female participants of childbearing potential must not be pregnant or breast-feeding, have a negative pregnancy test at screening and must be willing to undergo pregnancy testing throughout the study.
8. Both female participants of childbearing potential and male participants able to father a child must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two effective methods of contraception throughout the course of the study and for six weeks after the last investigational product injection. Acceptable methods of contraception for this study include:

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

1. Participant has a significant active infection (an infection requiring treatment as determined by the medical team), including active tuberculosis or human immunodeficiency virus (HIV).
2. Participant received a live vaccination within the past six weeks.
3. Participant is expected to receive a live vaccination at any time during the study.
4. Participant received the Bacillus Calmette-Guerin (BCG) vaccine within the past year.
5. Participant is expected to receive the BCG vaccine at any time during the study or up to one year after discontinuing ustekinumab.
6. Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years.
7. Participant has received intraocular (or periocular) steroid or anti-vascular endothelial growth factor (VEGF) injections within the last six weeks.
8. Participant received rituximab within the last six months or another biologic agent (e.g., infliximab, daclizumab, adalimumab) within the last two months.
9. Participant has received alkylating agents (e.g., cyclophosphamide, chlorambucil) within the last nine months.
10. Participant has a known hypersensitivity to ustekinumab or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-EI-0169.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Started | 5 | 3
Completed | 4 | 2
Not Completed | 1 | 1
Not completed — Insufficient Therapeutic Response | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous) | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9) | 48 (9) | 50 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Treatment Response by Week 16
Description: The primary outcome is the number of participants in each cohort who experience a treatment response by Week 16. Treatment response is defined as experiencing all of the following for both/eligible eyes: no active inflammatory chorioretinal lesion and/or absent or decreased retinal vascular leakage; ≤ 0.5+ anterior chamber (AC) cells; ≤ 0.5+ vitreous haze.
Time Frame: Baseline to Week 16
Population: All enrolled participants who received at least one dose of Ustekinumab and completed the Week 16 visit. One participant in each cohort is excluded from the analysis as a result of discontinuing the study prior to Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

2. Secondary Outcome: Mean Change in Visual Acuity in the Right Eye at All Follow-up Visits Compared to Baseline
Description: Mean change in visual acuity in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline as measured by electronic visual acuity (EVA).
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: All enrolled participants who received at least one dose of Ustekinumab and completed the Week 16 visit. One participant in each cohort is excluded from the analysis as a result of discontinuing the study prior to Week 16. At Week 28, one additional participant in Cohort 2 is excluded from the analysis due to missing visual acuity data.
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
letters read
  Week 4 | -1 (3) | -1 (1)
  Week 8 | 1 (3) | 1 (4)
  Week 12 | 2 (4) | 0 (3)
  Week 16 | 1 (8) | 0 (1)
  Week 28: number analyzed (Participants) | 4 | 1
  Week 28 | -2 (7) | -1 (NA) — Only one participant was analyzed for Cohort 2 at Week 28, so the standard deviation could not be calculated.

3. Secondary Outcome: Mean Change in Visual Acuity in the Left Eye at All Follow-up Visits Compared to Baseline
Description: Mean change in visual acuity in the left eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline as measured by electronic visual acuity (EVA).
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters read
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
letters read
  Week 4 | -2 (7) | 1 (4)
  Week 8 | 4 (5) | 1 (2)
  Week 12 | 4 (6) | 1 (2)
  Week 16 | 0 (13) | 0 (0)
  Week 28: number analyzed (Participants) | 4 | 1
  Week 28 | 6 (10) | -5 (NA) — Only one participant was analyzed for Cohort 2 at Week 28, so the standard deviation could not be calculated.

4. Secondary Outcome: Median Change in Visual Acuity in the Right Eye at All Follow-up Visits Compared to Baseline
Description: Median change in visual acuity in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline as measured by electronic visual acuity (EVA).
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 2
Measure: Median (Full Range); unit: letters read
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
letters read
  Week 4 | -1 [-4 to 2] | -1 [-1 to 0]
  Week 8 | 2 [-3 to 3] | 1 [-2 to 3]
  Week 12 | 3 [-2 to 5] | 0 [-2 to 2]
  Week 16 | 4 [-10 to 7] | 0 [-1 to 1]
  Week 28: number analyzed (Participants) | 4 | 1
  Week 28 | 1 [-12 to 4] | -1 [-1 to -1]

5. Secondary Outcome: Median Change in Visual Acuity in the Left Eye at All Follow-up Visits Compared to Baseline
Description: Median change in visual acuity in the left eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline as measured by electronic visual acuity (EVA).
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 2
Measure: Median (Full Range); unit: letters read
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
letters read
  Week 4 | -2 [-9 to 5] | 1 [-2 to 4]
  Week 8 | 2 [-1 to 11] | 1 [-1 to 2]
  Week 12 | 3 [-3 to 12] | 1 [-1 to 2]
  Week 16 | 1 [-16 to 15] | 0 [0 to 0]
  Week 28: number analyzed (Participants) | 4 | 1
  Week 28 | 3 [-3 to 20] | -5 [-5 to -5]

6. Secondary Outcome: Number of Participants Who Experience a Recurrence of Uveitis at All Follow-up Visits
Description: Number of participants in each cohort who experience a recurrence of uveitis at each follow-up visit (Week 4, Week 8, Week 12, and Week 16). Recurrence of uveitis is defined as the presence of one of the following in at least one eye: 1) new active inflammatory chorioretinal lesion and/or retinal vascular leakage; 2) a 2+ increase in anterior chamber (AC) cells relative to Baseline; 3) a 2-step increase in vitreous haze (VH) relative to Baseline; 4) worsening of best-corrected visual acuity (BCVA) by ≥ 15 letters relative to Baseline.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 0
  Week 16 | 1 | 0

7. Secondary Outcome: Mean Number of Days Until First Recurrence
Description: Mean number of days following the baseline injection until first recurrence (of the participants who recur). Recurrence of uveitis is defined as the presence of one of the following in at least one eye: 1) new active inflammatory chorioretinal lesion and/or retinal vascular leakage; 2) a 2+ increase in anterior chamber (AC) cells relative to Baseline; 3) a 2-step increase in vitreous haze (VH) relative to Baseline; 4) worsening of best-corrected visual acuity (BCVA) by ≥ 15 letters relative to Baseline.
Time Frame: Baseline to Week 16
Population: All enrolled participants who received at least one dose of Ustekinumab, completed the Week 16 visit, and experienced recurrence of uveitis. As only one participant experienced recurrence of uveitis, only one participant from Cohort 1 is included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 1 | 0
days | 118 (NA) — There was only participant analyzed for Cohort 1, so the standard deviation could not be calculated. |

8. Secondary Outcome: Median Number of Days Until First Recurrence
Description: Median number of days following the baseline injection until first recurrence (of the participants who recur). Recurrence of uveitis is defined as the presence of one of the following in at least one eye: 1) new active inflammatory chorioretinal lesion and/or retinal vascular leakage; 2) a 2+ increase in anterior chamber (AC) cells relative to Baseline; 3) a 2-step increase in vitreous haze (VH) relative to Baseline; 4) worsening of best-corrected visual acuity (BCVA) by ≥ 15 letters relative to Baseline.
Time Frame: Baseline to Week 16
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 1 | 0
days | 118 [118 to 118] |

9. Secondary Outcome: Presence or Extent of Macular Edema as Determined by Optical Coherence Tomography (OCT) in the Right Eye at All Follow-up Visits
Description: Presence or extent of macular edema as determined by optical coherence tomography (OCT) in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28). The number of participants that did and did not have macular edema present is presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: Present | 2 | 0
  Week 4: Not Present | 2 | 2
  Week 8: Present | 2 | 0
  Week 8: Not Present | 2 | 2
  Week 12: Present | 1 | 0
  Week 12: Not Present | 3 | 2
  Week 16: Present | 1 | 0
  Week 16: Not Present | 3 | 2
  Week 28: Present | 3 | 0
  Week 28: Not Present | 1 | 2

10. Secondary Outcome: Presence or Extent of Macular Edema as Determined by Optical Coherence Tomography (OCT) in the Left Eye at All Follow-up Visits
Description: Presence or extent of macular edema as determined by optical coherence tomography (OCT) in the left eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28). The number of participants that did and did not have macular edema present is presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: number analyzed (Participants) | 3 | 2
  Week 4: Present | 0 | 0
  Week 4: Not Present | 3 | 2
  Week 8: Present | 1 | 0
  Week 8: Not Present | 3 | 2
  Week 12: Present | 1 | 0
  Week 12: Not Present | 3 | 2
  Week 16: Present | 1 | 0
  Week 16: Not Present | 3 | 2
  Week 28: Present | 2 | 0
  Week 28: Not Present | 2 | 2

11. Secondary Outcome: Presence or Extent of Macular Edema as Determined by Fluorescein Angiogram (FA) in the Right Eye at All Follow-up Visits
Description: Presence or extent of macular edema as determined by fluorescein angiogram (FA) in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28). The number of participants that did and did not have macular edema present is presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: All enrolled participants who received at least one dose of Ustekinumab and completed the Week 16 visit. One participant in each cohort is excluded from the analysis as a result of discontinuing the study prior to Week 16. No participants in Cohort 2 were analyzed at Week 4 as neither had FA performed at that visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: number analyzed (Participants) | 2 | 0
  Week 4: Present | 2 |
  Week 4: Not Present | 0 |
  Week 8: Present | 4 | 0
  Week 8: Not Present | 0 | 2
  Week 12: number analyzed (Participants) | 3 | 2
  Week 12: Present | 3 | 0
  Week 12: Not Present | 0 | 2
  Week 16: Present | 3 | 0
  Week 16: Not Present | 1 | 2
  Week 28: Present | 3 | 1
  Week 28: Not Present | 1 | 1

12. Secondary Outcome: Presence or Extent of Macular Edema as Determined by Fluorescein Angiogram (FA) in the Left Eye at All Follow-up Visits
Description: Presence or extent of macular edema as determined by fluorescein angiogram (FA) in the left eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28). The number of participants that did and did not have macular edema present is presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: number analyzed (Participants) | 2 | 0
  Week 4: Present | 1 |
  Week 4: Not Present | 1 |
  Week 8: Present | 2 | 0
  Week 8: Not Present | 2 | 2
  Week 12: number analyzed (Participants) | 3 | 2
  Week 12: Present | 3 | 0
  Week 12: Not Present | 0 | 2
  Week 16: Present | 3 | 1
  Week 16: Not Present | 1 | 1
  Week 28: Present | 4 | 2
  Week 28: Not Present | 0 | 0

13. Secondary Outcome: Amount of Retino-vascular Leakage as Measured by Fluorescein Angiogram (FA) in the Right Eye at All Follow-up Visits
Description: Amount of retino-vascular leakage as measured by fluorescein angiogram (FA) in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28). The number of participants experiencing presence and new/increased lesions, presence and decreased lesions, presence and no new/increased or decreased lesions, and absence of lesions are presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: Presence and New/Increased Lesions | 0 | 0
  Week 4: Presence and Decreased Lesions | 0 | 0
  Week 4: Presence and No New/Increased or Decreased Lesions | 1 | 0
  Week 4: Absence of Lesions | 3 | 2
  Week 8: Presence and New/Increased Lesions | 0 | 0
  Week 8: Presence and Decreased Lesions | 0 | 0
  Week 8: Presence and No New/Increased or Decreased Lesions | 0 | 1
  Week 8: Absence of Lesions | 4 | 1
  Week 12: Presence and New/Increased Lesions | 0 | 0
  Week 12: Presence and Decreased Lesions | 0 | 0
  Week 12: Presence and No New/Increased or Decreased Lesions | 0 | 2
  Week 12: Absence of Lesions | 4 | 0
  Week 16: Presence and New/Increased Lesions | 1 | 0
  Week 16: Presence and Decreased Lesions | 0 | 0
  Week 16: Presence and No New/Increased or Decreased Lesions | 0 | 1
  Week 16: Absence of Lesions | 3 | 1
  Week 28: Presence and New/Increased Lesions | 0 | 0
  Week 28: Presence and Decreased Lesions | 0 | 0
  Week 28: Presence and No New/Increased or Decreased Lesions | 0 | 0
  Week 28: Absence of Lesions | 4 | 2

14. Secondary Outcome: Amount of Retino-vascular Leakage as Measured by Fluorescein Angiogram (FA) in the Left Eye at All Follow-up Visits
Description: Amount of retino-vascular leakage as measured by fluorescein angiogram (FA) in the left eye at all follow-up visits (Week 4, week 8, Week 12, Week 16, and Week 28). The number of participants experiencing presence and new/increased lesions, presence and decreased lesions, presence and no new/increased or decreased lesions, and absence of lesions are presented.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants
  Week 4: Presence and New/Increased Lesions | 0 | 0
  Week 4: Presence and Decreased Lesions | 0 | 0
  Week 4: Presence and No New/Increased or Decreased Lesions | 1 | 0
  Week 4: Absence of Lesions | 3 | 2
  Week 8: Presence and New/Increased Lesions | 0 | 0
  Week 8: Presence and Decreased Lesions | 0 | 0
  Week 8: Presence and No New/Increased or Decreased Lesions | 0 | 0
  Week 8: Absence of Lesions | 4 | 2
  Week 12: Presence and New/Increased Lesions | 0 | 0
  Week 12: Presence and Decreased Lesions | 0 | 0
  Week 12: Presence and No New/Increased or Decreased Lesions | 0 | 1
  Week 12: Absence of Lesions | 4 | 1
  Week 16: Presence and New/Increased Lesions | 1 | 0
  Week 16: Presence and Decreased Lesions | 0 | 0
  Week 16: Presence and No New/Increased or Decreased Lesions | 0 | 0
  Week 16: Absence of Lesions | 3 | 2
  Week 28: Presence and New/Increased Lesions | 0 | 0
  Week 28: Presence and Decreased Lesions | 0 | 0
  Week 28: Presence and No New/Increased or Decreased Lesions | 0 | 0
  Week 28: Absence of Lesions | 4 | 2

15. Secondary Outcome: Changes in Central Retinal Thickness as Measured by Optical Coherence Tomography (OCT) in the Right Eye at All Follow-up Visits Compared to Baseline
Description: Mean change in central retinal thickness as measured by optical coherence tomography (OCT) in the right eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline.
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
micrometers
  Week 4 | 8 (14) | -2 (4)
  Week 8 | -49 (95) | -6 (12)
  Week 12 | -11 (13) | 6 (1)
  Week 16 | -28 (16) | -7 (16)
  Week 28 | -9 (40) | -2 (11)

16. Secondary Outcome: Changes in Central Retinal Thickness as Measured by Optical Coherence Tomography (OCT) in the Left Eye at All Follow-up Visits Compared to Baseline
Description: Mean change in central retinal thickness as measured by optical coherence tomography (OCT) in the left eye at all follow-up visits (Week 4, Week 8, Week 12, Week 16, and Week 28) compared to baseline.
Time Frame: Baseline to Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
micrometers
  Week 4 | -13 (26) | 1 (1)
  Week 8 | 17 (34) | -1 (6)
  Week 12 | 54 (87) | 2 (4)
  Week 16 | -2 (31) | 8 (6)
  Week 28 | -1 (24) | 19 (6)

17. Secondary Outcome: Length of Time to Quiescence in the Right Eye
Description: Mean length of time to first experience of quiescence in the right eye. Quiescence refers to absence of active disease defined as not having the following conditions: +1 or more vitreous haze; and/or active chorioretinitis or leakage on fluorescein angiogram (FA) (that is more than one quadrant) that requires treatment.
Time Frame: Baseline to Week 16
Population: All enrolled participants who received at least one dose of Ustekinumab, completed the Week 16 visit, and experienced quiescence. One participant in each cohort is excluded from the analysis as a result of discontinuing the study prior to Week 16. An additional participant in Cohort 1 is excluded due to not experiencing quiescence.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 3 | 2
days | 24 (8) | 38 (8)

18. Secondary Outcome: Length of Time to Quiescence in the Left Eye
Description: Mean length of time to first experience of quiescence in the left eye. Quiescence refers to absence of active disease defined as not having the following conditions: +1 or more vitreous haze; and/or active chorioretinitis or leakage on fluorescein angiogram (FA) (that is more than one quadrant) that requires treatment.
Time Frame: Baseline to Week 16
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 3 | 2
days | 38 (16) | 38 (8)

19. Secondary Outcome: Ability to Taper Concomitant Immunosuppressive Medications
Description: The number of participants able to taper concomitant immunosuppressive medications.
Time Frame: Baseline to Week 28
Population: All enrolled participants who received at least one dose of Ustekinumab and completed the Week 16 visit. One participant in Cohort 1 is excluded from the analysis as a result of discontinuing the study prior to Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants | 1 | 0

20. Other Pre Specified Outcome: Number of Participants Experiencing a Clinically Significant Increase in Elevated Intraocular Pressure (IOP) at Any Follow-up Visit
Description: Number of participants experiencing a clinically significant increase in elevated intraocular pressure (IOP) at any follow-up visit in either eye. An increase in IOP ≥10 mmHg as compared with baseline is considered a clinically significant increase.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants | 2 | 0

21. Other Pre Specified Outcome: Proportion of Participants With ≥15 Letter Loss at Any Follow-up Visit.
Description: Proportion of participants with ≥15 letter loss in best-corrected visual acuity (BCVA) from baseline at any follow-up visit in either eye.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
Participants | 1 | 0

22. Other Pre Specified Outcome: Number and Severity of Systemic and Ocular Toxicities and Adverse Events
Description: Number and severity of systemic and ocular toxicities and adverse events for participants in both cohorts. Severity of each event is classified as mild, moderate, or severe. Natural progression of disease adverse events are not included.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Number; unit: adverse events
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
Number analyzed (Participants) | 4 | 2
adverse events
  Mild | 10 | 7
  Moderate | 3 | 3
  Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Cohort 1 (Subcutaneous Only) | Cohort 2 (IV and Subcutaneous)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Subcutaneous Only) (N=5) | Cohort 2 (IV and Subcutaneous) (N=3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) — Natural progression of disease event
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) — Natural progression of disease event
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) — Natural progression of disease event
Subretinal fluid (Eye disorders) | 1 (1) | 0 (0) — Natural progression of disease event
Cystoid macular oedema (Eye disorders) | 1 (2) | 0 (0) — Natural progression of disease event
Iris adhesions (Eye disorders) | 1 (1) | 0 (0) — Natural progression of disease event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02911116/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT02911116/SAP_001.pdf